CLINICAL TRIAL: NCT04255589
Title: A Phase 3, Multi-center, Randomized, Double-blind, Parallel-group Trial to Evaluate the Efficacy and Safety of CKD-495 in Patients With Acute and Chronic Gastritis
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of CKD-495
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A74_02AG/CG1904
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Gastritis
Keywords: Acute Gastritis; Chronic Gastritis; Cinnamic acid; CKD-495
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients assigned to this group are treated with one CKD-495 75mg Tab.,and one Placebo Tab.(Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg Tab)
  Interventions: Drug: CKD-495 75mg; Drug: Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg
- Active comparator Group (Active Comparator): Patients assigned to this group are treated with one Artemisiae argyi folium 95% ethanol ext.(20→1) 60mg Tab, and one Placebo Tab.(Placebo of the CKD-495 75mg)
  Interventions: Drug: Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg; Drug: Placebo of the CKD-495 75mg

INTERVENTIONS:
Drug: CKD-495 75mg — CKD-495 75mg Tab.
  Arms: Experimental Group
Drug: Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg — Artemisiae argyi folium 95% ethanol ext.(20→1) 60mg Tab.
  Arms: Active comparator Group
Drug: Placebo of the CKD-495 75mg — Placebo of the CKD-495 75mg Tab.
  Arms: Active comparator Group
Drug: Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg — Placebo of Artemisia Herb 95% Ethanol Soft Ext.(20→1) 60mg Tab.
  Arms: Experimental Group

SUMMARY:
To Evaluate the Efficacy and Safety of CKD-495

DETAILED DESCRIPTION:
A phase 3, Multi-center, Randomized, Double-blind, Parallel-group Trial to Evaluate the Efficacy and Safety of CKD-495 in Patients With Acute and Chronic Gastritis

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subjects aged ≥ 19
2. Acute or Chronic gastritis patients who have more than 1 erosion on endoscopy within 7days prior to the use of the Investigator's Product taken date
3. Patients who have more than 1 subjective symptom

Exclusion Criteria:

1. Patients with peptic ulcer, gastroesophageal reflux disease, malignant tumor in the digestive system or coagulation disorder, or taking antithrombotic medicine
2. Patients who have been taken any gastritis medicine that could affect the treatment: H2 receptor antagonist, PPI(Proton Pump Inhibitor), antacid, improvement of movement in digestive system, Prostaglandin, and protective agent for gastritis
3. Patients who have to take medicine that could cause gastritis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Improvement rate of gastric erosion | 14days after drug administrations
  50% change on erosive grade

SECONDARY OUTCOMES:
cure rate of gastric erosion | 14days after drug administrations
  0 erosion
Improvement rate of symptoms | 14days after drug administrations
  50% change on the Subjective Symptoms total score
Improvement rate of gastric edema | 14days after drug administrations
  50% change on the Edema grade
Improvement rate of gastric erythema | 14days after drug administrations
  50% change on the Erythema grade
Improvement rate of gastric hemorrhage | 14days after drug administrations
  50% change on the Hemorrhage grade

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Lee, MD, Ph.D., Principal Investigator — Hanyang University
Locations (17):
- South Korea (17):
  - Chonnam National University Hospital, Gwangju, Donggu
  - Kyoungpook National University Hospital, Daegu, Gyeongsangbuk-do
  - Busan National University Hospital, Busan, Seo-gu
  - Inje University Busan Paik Hospital, Busan
  - Yeungnam University Medical Center, Daegu
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam
  - Chung Ang University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Yeouido ST. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seo SY, Lee ST, Kim SK, Chun HJ, Song GA, Lee DH, Kim JJ, Kim JI, Lee YC, Kim TN, Jee SR, Park SY, Kim JG, Park JJ, Kim SG, Park JM, Park JH, Park SJ, Lee OY. Efficacy and safety of CKD-495 in acute and chronic gastritis: A Phase III superiority clinical trial. Medicine (Baltimore). 2023 Dec 8;102(49):e35926. doi: 10.1097/MD.0000000000035926. PMID 38065906